CLINICAL TRIAL: NCT02717767
Title: Measuring Auto-fluorescence of White Corpuscles for the Early Diagnosis and the Monitoring of Pneumonia in Intensive Care Units
Brief Title: Measuring Auto-fluorescence of White Corpuscles for the Early Diagnosis and the Monitoring of Pneumonia in ICU
Acronym: BIONAGA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0081
Record Dates: First submitted 2016-03-14; First posted 2016-03-24 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Pneumonia
Keywords: pneumonia; diagnosis; prognosis; tracheal aspirate; bronchoalveolar lavage
MeSH Terms: conditions — Pneumonia; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tracheal aspirate and bronchoalveolar lavages
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Autofluorescence of white corpuscle — Measure of auto-fluorescence of white corpuscles cells harvested from tracheal aspirate and/or bronchoalveolar lavages

SUMMARY:
The diagnosis of pneumonia is challenging in Intensive Care Unit. The auto-fluorescence of white corpuscles is altered during pneumonia. In presence of bacterial growth on lung samples, the measure of autofluorescence of white corpuscles could help the clinicians to discriminate bacterial colonization from acute infection.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in intensive care units
* Mechanical ventilation
* Age > 18 years
* Collection of a lung sample for bacteriological analysis for the suspicion of a first episode of lung infection.

Exclusion Criteria:

* Refuse to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04-21 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Pneumonia | 28 days
  Diagnosis of pneumonia (Clinical Pulmonary Infection Score > 6, with assessment of the chest radiography by a blinded investigator)

SECONDARY OUTCOMES:
Clinical Pulmonary Infection Score > 6 | day 3
Acute respiratory distress syndrome | day 90
  PaO2/FiO2 < 200 with a PEEP > 5 (Berlin definition)
Duration of mechanical ventilation | day 90
Intensive Care unit Length of stay | day 90
Mortality | day 90

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ROQUILLY, PH, Principal Investigator — Nantes University Hospital
Locations (4):
- France (4):
  - Blois Hospital, Blois
  - Saint-Brieuc Hospital, Saint-Brieuc
  - Saint-NazaireHospital, Saint-Nazaire
  - Vannes Hospital, Vannes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monsel A, Lecart S, Roquilly A, Broquet A, Jacqueline C, Mirault T, Troude T, Fontaine-Aupart MP, Asehnoune K. Analysis of autofluorescence in polymorphonuclear neutrophils: a new tool for early infection diagnosis. PLoS One. 2014 Mar 21;9(3):e92564. doi: 10.1371/journal.pone.0092564. eCollection 2014. PMID 24658436